CLINICAL TRIAL: NCT03575871
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, MULTI-CENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PF-04965842 MONOTHERAPY IN SUBJECTS AGED 12 YEARS AND OLDER, WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Study Evaluating Efficacy and Safety of PF-04965842 in Subjects Aged 12 Years And Older With Moderate to Severe Atopic Dermatitis
Acronym: JADE Mono-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451013; MONO-2 (Other: Alias Study Number); 2018-001136-21 (EudraCT Number)
Record Dates: First submitted 2018-06-15; First posted 2018-07-03 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-04965842 100 mg (Experimental)
  Interventions: Drug: PF-04965842 100 mg
- PF-04965842 200 mg (Experimental)
  Interventions: Drug: PF-04965842 200 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 100 mg — PF-04965842 100 mg, administered as two tablets to be taken orally once daily for 12 weeks
  Arms: PF-04965842 100 mg
Drug: PF-04965842 200 mg — PF-04965842 200 mg, administered as two tablets to be taken orally once daily for 12 weeks
  Arms: PF-04965842 200 mg
Drug: Placebo — Placebo, administered as two tablets to be taken orally once daily for 12 weeks
  Arms: Placebo

SUMMARY:
B7451013 is a Phase 3 study to evaluate PF-04965842 in patients aged 12 years and older with a minimum body weight of 40 kg who have moderate to severe atopic dermatitis. The efficacy and safety of two dosage strengths of PF-04965842, 100 mg and 200 mg taken orally once daily, will be evaluated relative to placebo over 12 weeks of study participation. Eligible patients will have an option to enter a long-term extension study after completing 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older with a minimum body weight of 40 kg
* Diagnosis of atopic dermatitis (AD) for at least 1 year and current status of moderate to severe disease (>= the following scores: BSA 10%, IGA 3, EASI 16, Pruritus NRS severity 4)
* Recent history of inadequate response or inability to tolerate topical AD treatments or require systemic treatments for AD control

Exclusion Criteria:

* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
* Prior treatment with JAK inhibitors
* Other active nonAD inflammatory skin diseases or conditions affecting skin
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use contraception

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (115):
- United States (28):
  - Emmaus Research Center, Inc., Anaheim, California
  - Advanced Research Center, Inc. - Los Alamitos Site, Los Alamitos, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Clinical Science Institute, Santa Monica, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Colorado Springs Dermatology Clinic, PC, Colorado Springs, Colorado
  - Olympian Clinical Research, Clearwater, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Precision Imaging, Jacksonville, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Imaging Center of Idaho, Caldwell, Idaho
  - ASR, LLC, Nampa, Idaho
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Sadick Research Group, New York, New York
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Ohio State University Dermatology East, Gahanna, Ohio
  - Tanenbaum Dermatology Center, Memphis, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Austin Institute for Clinical Research, Inc. - Central, Austin, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - West Houston Dermatology, PA, Houston, Texas
  - Summit Clinical Research, LLC, Franklin, Virginia
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Australia (7):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Skin and Cancer Foundation Inc, Carlton, VIC 3053
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Royal Children's Hospital (RCH), Parkville, Victoria
- Bulgaria (6):
  - Medical Centre Asklepii OOD, Dupnitsa
  - MHAT Dr. Tota Venkova AD, Gabrovo
  - "Acibadem City Clinic MHAT Tokuda" EAD, Sofia
  - "DCC Aleksandrovska" EOOD, Sofia
  - Diagnostic Consultative Center Fokus-5, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
- Canada (7):
  - University of British Columbia Department of Dermatology and Skin Science, Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - North York Research Inc., North York, Ontario
  - Oshawa Clinic Dermatology Trials, Oshawa, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Army Medical University, PLA, Chongqing, Chongqing Municipality
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Tianjin Medical University General Hospital, Dermatological Department, Tianjin
- Czechia (7):
  - Dermamedica S.R.O., Náchod
  - Oblastni nemocnice Nachod a.s., Radiodiagnosticke oddeleni, Náchod
  - Lekarna u Stribrneho orla, Náchod
  - Sanatorium profesora Arenbergera, Prague
  - Lekarna U sv. Ignace, Prague
  - Dermatologicka Ambulance, Svitavy
  - Lekarna na Hranicni, Svitavy
- Germany (7):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - ISA GmbH, Berlin
  - Fachärztliche Gemeinschaftspraxis für Dermatologie und Venerologie, Allergologie,, Blankenfelde-Mahlow
  - IKF Pneumologie GmbH & Co KG, Frankfurt
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Universitaet Muenster, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (4):
  - SE AOK Bor, Nemikortani es Boronkologiai Klinika, Budapest
  - Budapest Főváros XIX. Kerületi Önkormányzat Kispesti Egészsegügyi Intézete, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - ALLERGO-DERM BAKOS Kft., Szolnok
- Japan (8):
  - Queen's square Medical Facilities Queen's square Dermatology and Allergology, Yokohama, Kanagawa
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Kume Clinic, Sakai, Osaka
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - Matsuyama Dermatology Clinic, Nakano-ku, Tokyo
  - Hoshikuma Dermatology・Allergy Clinic, Fukuoka
  - Sanrui Hifuka, Saitama
- Latvia (5):
  - Selga Freiberga private practice in dermatovenerology and cosmetology, Jelgava
  - Riga 1st Hospital, Clinic for Dermatology and STD, Riga
  - Aesthetic dermatology clinic of Prof. J. Kisis, Riga
  - Health Centre 4 Ltd. Diagnostics Centre, Riga
  - Health Centre 4 Ltd, Riga
- Poland (15):
  - NZOZ Specjalistyczny Osrodek Dermatologiczny DERMAL s.c., Bialystok
  - KLIMED Marek Klimkiewicz, Bialystok
  - Centrum Badań Klinicznych JCI, Krakow
  - Centrum Nowoczesnych Terapii "DOBRY LEKARZ" sp. z o. o., Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Clinical Research Center Sp. z o.o. MEDIC-R Sp. k., Poznan
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Synexus Polska Sp. z o. o. Oddzial w Warszawie, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Klinika Ambroziak Sp. z o.o., Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - Lukasz Matusiak "4HEALTH", Wroclaw
- South Korea (10):
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Bupyeong-gu, Incheon
  - Inha University Hospital, Jung-gu, Incheon
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei Univ. Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym university Kangnam Sacred Heart Hospital, Seoul
- United Kingdom (6):
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth, Devon
  - MAC Clinical Research, Blackpool, Lancashire
  - MAC Clinical Research Ltd, Cannock, South Staffordshire
  - Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - MAC Clinical Research Ltd, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Paller AS, Eichenfield LF, Irvine AD, Flohr C, Wollenberg A, Barbarot S, Bangert C, Spergel JM, Selfridge A, Biswas P, Fan H, Alderfer J, Watkins M, Koppensteiner H. Integrated Efficacy and Safety Analysis of Abrocitinib in Adolescents With Moderate-to-Severe Atopic Dermatitis. Allergy. 2025 Aug;80(8):2213-2224. doi: 10.1111/all.16512. Epub 2025 Mar 3. PMID 40028832
- [Derived] Silverberg JI, Thyssen JP, Lazariciu I, Myers DE, Guler E, Chovatiya R. Abrocitinib may improve itch and quality of life in patients with itch-dominant atopic dermatitis. Skin Health Dis. 2024 May 5;4(4):e382. doi: 10.1002/ski2.382. eCollection 2024 Aug. PMID 39104653
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Schmid-Grendelmeier P, Gooderham MJ, Hartmann K, Konstantinou GN, Fellmann M, Koulias C, Clibborn C, Biswas P, Brunner PM. Efficacy and safety of abrocitinib in patients with moderate-to-severe atopic dermatitis and comorbid allergies. Allergy. 2024 Jan;79(1):174-183. doi: 10.1111/all.15952. Epub 2023 Nov 21. PMID 37988255
- [Derived] Alexis AF, Silverberg JI, Rice ZP, Armstrong AW, Desai SR, Fonacier L, Kabashima K, Biswas P, Cella RR, Chan GL, Levenberg M. Abrocitinib efficacy and safety in moderate-to-severe atopic dermatitis by race, ethnicity, and Fitzpatrick skin type. Ann Allergy Asthma Immunol. 2024 Mar;132(3):383-389.e3. doi: 10.1016/j.anai.2023.11.002. Epub 2023 Nov 10. PMID 37949351
- [Derived] Yosipovitch G, Gooderham MJ, Stander S, Fonacier L, Szepietowski JC, Deleuran M, Girolomoni G, Su JC, Bushmakin AG, Cappelleri JC, Feeney C, Chan G, Thorpe AJ, Valdez H, Biswas P, Rojo R, DiBonaventura M, Myers DE. Interpreting the Relationship Among Itch, Sleep, and Work Productivity in Patients with Moderate-to-Severe Atopic Dermatitis: A Post Hoc Analysis of JADE MONO-2. Am J Clin Dermatol. 2024 Jan;25(1):127-138. doi: 10.1007/s40257-023-00810-7. Epub 2023 Aug 25. PMID 37624488
- [Derived] Blauvelt A, Boguniewicz M, Brunner PM, Luna PC, Biswas P, DiBonaventura M, Farooqui SA, Rojo R, Cameron MC. Abrocitinib monotherapy in Investigator's Global Assessment nonresponders: improvement in signs and symptoms of atopic dermatitis and quality of life. J Dermatolog Treat. 2022 Aug;33(5):2605-2613. doi: 10.1080/09546634.2022.2059053. Epub 2022 Jul 6. PMID 35763326
- [Derived] Stander S, Bhatia N, Gooderham MJ, Silverberg JI, Thyssen JP, Biswas P, DiBonaventura M, Romero W, Farooqui SA. High threshold efficacy responses in moderate-to-severe atopic dermatitis are associated with additional quality of life benefits: pooled analyses of abrocitinib monotherapy studies in adults and adolescents. J Eur Acad Dermatol Venereol. 2022 Aug;36(8):1308-1317. doi: 10.1111/jdv.18170. Epub 2022 May 6. PMID 35462428
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population pharmacokinetic-pharmacodynamic modelling of platelet time-courses following administration of abrocitinib. Br J Clin Pharmacol. 2022 Aug;88(8):3856-3871. doi: 10.1111/bcp.15334. Epub 2022 Apr 11. PMID 35342978
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- [Derived] Cork MJ, McMichael A, Teng J, Valdez H, Rojo R, Chan G, Zhang F, Myers DE, DiBonaventura M. Impact of oral abrocitinib on signs, symptoms and quality of life among adolescents with moderate-to-severe atopic dermatitis: an analysis of patient-reported outcomes. J Eur Acad Dermatol Venereol. 2022 Mar;36(3):422-433. doi: 10.1111/jdv.17792. Epub 2021 Dec 4. PMID 34743361
- [Derived] Simpson EL, Silverberg JI, Nosbaum A, Winthrop KL, Guttman-Yassky E, Hoffmeister KM, Egeberg A, Valdez H, Zhang M, Farooqui SA, Romero W, Thorpe AJ, Rojo R, Johnson S. Integrated Safety Analysis of Abrocitinib for the Treatment of Moderate-to-Severe Atopic Dermatitis From the Phase II and Phase III Clinical Trial Program. Am J Clin Dermatol. 2021 Sep;22(5):693-707. doi: 10.1007/s40257-021-00618-3. Epub 2021 Aug 18. PMID 34406619
- [Derived] Silverberg JI, Thyssen JP, Simpson EL, Yosipovitch G, Stander S, Valdez H, Rojo R, Biswas P, Myers DE, Feeney C, DiBonaventura M. Impact of Oral Abrocitinib Monotherapy on Patient-Reported Symptoms and Quality of Life in Adolescents and Adults with Moderate-to-Severe Atopic Dermatitis: A Pooled Analysis of Patient-Reported Outcomes. Am J Clin Dermatol. 2021 Jul;22(4):541-554. doi: 10.1007/s40257-021-00604-9. Epub 2021 May 5. PMID 33954933
- [Derived] Silverberg JI, Simpson EL, Thyssen JP, Gooderham M, Chan G, Feeney C, Biswas P, Valdez H, DiBonaventura M, Nduaka C, Rojo R. Efficacy and Safety of Abrocitinib in Patients With Moderate-to-Severe Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2020 Aug 1;156(8):863-873. doi: 10.1001/jamadermatol.2020.1406. PMID 32492087
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with age greater than or equal to (>=) 12 years with moderate to severe atopic dermatitis (AD) and a body weight of >=40 kilograms were enrolled in the study. Eligible participants had an option to enter into a long-term extension (LTE) study after completing 12 weeks of treatment in this study.
Pre-assignment Details: This study was conducted from 29-June-2018 to 13-Aug-2019 at 106 sites in 13 countries.
Groups:
- PF-04965842 100 mg: Participants were randomized to receive a tablet of PF-04965842 (abrocitinib) 100 milligrams (mg) and a tablet of matching placebo orally once daily for 12 weeks. Participants who discontinued early from treatment or who were not eligible for LTE study, were followed up to 4 weeks after last dose of study drug.
- PF-04965842 200 mg: Participants were randomized to receive PF-04965842 200 mg (2 tablets of 100 mg each) orally once daily for 12 weeks. Participants who discontinued early from treatment or who were not eligible for LTE study, were followed up to 4 weeks after last dose of study drug.
- Placebo: Participants were randomized to receive 2 tablets of placebo matched to PF-04965842 100 mg orally once daily for 12 weeks. Participants who discontinued early from treatment or who were not eligible for LTE study, were followed up to 4 weeks after last dose of study drug.
Period: Overall Study
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Started | 158 | 155 | 78
Completed | 137 | 141 | 52
Not Completed | 21 | 14 | 26
Not completed — Adverse Event | 5 | 5 | 8
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 4 | 7
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Protocol Deviation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 6 | 1 | 9
Not completed — Other than specified | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo | Total
Number analyzed (Participants) | 158 | 155 | 78 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (15.8) | 33.5 (14.7) | 33.4 (13.8) | 35.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 67 | 31 | 162
  Male | 94 | 88 | 47 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 2 | 9
  Not Hispanic or Latino | 154 | 150 | 73 | 377
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 46 | 54 | 29 | 129
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 6 | 21
  White | 101 | 91 | 40 | 232
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of Clear (0) or Almost Clear (1) and Greater Than or Equal to (>=) 2 Points Improvement From Baseline at Week 12
Description: IGA assesses severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Assessment excluded soles, palms and scalp.
Time Frame: Baseline, Week 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 155 | 155 | 77
percentage of participants | 28.4 [21.3 to 35.5] | 38.1 [30.4 to 45.7] | 9.1 [2.7 to 15.5]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; The estimate and confidence interval (CI) for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 19.3, 95% CI 2-sided [9.6 to 29.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 28.7, 95% CI 2-sided [18.6 to 38.8]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=75 Percent (%) Improvement (EASI-75) From Baseline at Week 12
Description: EASI evaluates severity of participants AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks] on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 155 | 154 | 77
percentage of participants | 44.5 [36.7 to 52.3] | 61.0 [53.3 to 68.7] | 10.4 [3.6 to 17.2]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.9, 95% CI 2-sided [23.3 to 44.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 50.5, 95% CI 2-sided [40.0 to 60.9]

3. Secondary Outcome: Percentage of Participants Who Achieved at Least 4-Points Improvement From Baseline in the Numerical Rating Scale (NRS) for Severity of Pruritus at Weeks 2, 4, 8 and 12
Description: Participants were asked to assess their worst pruritus/itching due to AD over the past 24 hours on an NRS scale ranged from 0 (no itching) to 10 (worst possible itching), where higher scores indicated greater severity.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 76
percentage of participants
  Week 2 | 23.1 [16.5 to 29.7] | 35.3 [27.7 to 42.9] | 3.9 [0.0 to 8.3]
  Week 4 | 31.4 [24.1 to 38.7] | 50.3 [42.4 to 58.2] | 3.9 [0.0 to 8.3]
  Week 8 | 39.1 [31.4 to 46.8] | 51.6 [43.7 to 59.6] | 11.8 [4.6 to 19.1]
  Week 12 | 39.7 [32.1 to 47.4] | 49.0 [41.1 to 56.9] | 10.5 [3.6 to 17.4]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Week 2: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 19.2, 95% CI 2-sided [11.0 to 27.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 31.2, 95% CI 2-sided [22.3 to 40.2]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; Week 4: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 27.5, 95% CI 2-sided [18.9 to 36.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 46.4, 95% CI 2-sided [37.2 to 55.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; Week 8: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 27.4, 95% CI 2-sided [16.8 to 38.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 39.8, 95% CI 2-sided [28.9 to 50.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; Week 12: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 29.3, 95% CI 2-sided [18.9 to 39.6]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 38.6, 95% CI 2-sided [28.1 to 49.1]

4. Secondary Outcome: Change From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis (PSAAD) Total Score at Week 12
Description: PSAAD is a daily participant reported symptom electronic diary. Participants rated their symptoms of AD over the past 24 hours, using 11 items (itchy skin, painful skin, dry skin, flaky skin, cracked skin, bumpy skin, red skin, discolored skin [lighter or darker], bleeding from skin, seeping or oozing fluid from skin [other than blood], and skin swelling). Participant had to think about all the areas of their body affected by their skin condition and chose the number that best described their experience for each of the 11 items, from 0 (no symptoms) to 10 (extreme symptoms), higher scores signified worse skin condition. Total PSAAD score = arithmetic mean of 11 items, 0 (no symptoms) to 10 (extreme symptoms), where higher score = worse skin condition.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 155 | 77
units on a scale | -2.4 [-2.8 to -2.1] | -3.0 [-3.3 to -2.7] | -0.8 [-1.3 to -0.3]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Mixed Model Repeated Measure (MMRM) contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category), baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.7, 95% CI 2-sided [-2.3 to -1.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.2, 95% CI 2-sided [-2.8 to -1.6]

5. Secondary Outcome: Time to Achieve >=4 Points Improvement From Baseline in Numerical Rating Scale (NRS) for Severity of Pruritus
Description: Participants were asked to assess their worst itching/pruritus due to AD over the past 24 hours on an NRS scale ranged from 0 (no itching) to 10 (worst itch imaginable), where higher scores indicated greater severity.
Time Frame: Baseline up to Day 15
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 90 | 110 | 20
days | 58.0 [11.0 to NA] — Upper limit was not evaluable as too few events were observed. | 29.0 [8.0 to 87.0] | 112.0 [58.0 to NA] — upper limit was not evaluable as too few events were observed.

6. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=75% Improvement (EASI-75) From Baseline at Weeks 2, 4 and 8
Description: EASI evaluates severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Number Analyzed" signifies the number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 10.2 [5.5 to 14.9] | 24.3 [17.5 to 31.2] | 1.3 [0.0 to 3.9]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 26.5 [19.5 to 33.4] | 51.0 [43.1 to 58.9] | 6.5 [1.0 to 12.0]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 43.3 [35.6 to 51.1] | 60.4 [52.7 to 68.1] | 12.8 [5.4 to 20.2]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0150, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 8.8, 95% CI 2-sided [2.8 to 14.9]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 22.7, 95% CI 2-sided [15.0 to 30.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.0, 95% CI 2-sided [10.9 to 29.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 44.3, 95% CI 2-sided [34.8 to 53.8]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 30.4, 95% CI 2-sided [19.7 to 41.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 47.4, 95% CI 2-sided [36.8 to 58.0]

7. Secondary Outcome: Percentage of Participants Achieving IGA Response of Clear (0) or Almost Clear (1) and >=2 Points Improvement From Baseline at Weeks 2, 4 and 8
Description: IGA assesses severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Assessment excluded sole, palms and scalp.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 5.1 [1.7 to 8.5] | 14.5 [8.9 to 20.1] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 14.2 [8.7 to 19.7] | 33.3 [25.9 to 40.8] | 1.3 [0.0 to 3.8]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 22.3 [15.8 to 28.8] | 37.7 [30.0 to 45.3] | 10.3 [3.5 to 17.0]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0459, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.1, 95% CI 2-sided [0.2 to 10.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 14.2, 95% CI 2-sided [7.8 to 20.5]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 12.9, 95% CI 2-sided [6.3 to 19.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 31.8, 95% CI 2-sided [23.6 to 39.9]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0246, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 11.9, 95% CI 2-sided [2.4 to 21.4]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 26.9, 95% CI 2-sided [17.0 to 36.9]

8. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of Clear (0) at Week 2, 4, 8 and 12
Description: as for outcome 1
Time Frame: Weeks 2, 4, 8 and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Number Analyzed" signifies number of participants evaluable at the specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 0 [0.0 to 2.3] | 2.0 [0.0 to 4.2] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 1.9 [0.0 to 4.1] | 4.6 [1.3 to 7.9] | 0 [0.0 to 4.7]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 1.3 [0.0 to 3.0] | 4.5 [1.3 to 7.8] | 0 [0.0 to 4.6]
  Week 12: number analyzed (Participants) | 155 | 155 | 77
  Week 12 | 5.2 [1.7 to 8.6] | 6.5 [2.6 to 10.3] | 0 [0.0 to 4.7]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; P-value was not estimable since there were no events; Difference in Percentage = 0.0, 95% CI 2-sided [-3.7 to 3.7]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2262, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.9, 95% CI 2-sided [-2.2 to 6.1]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.2223, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.9, 95% CI 2-sided [-2.2 to 6.1]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0597, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.5, 95% CI 2-sided [-0.2 to 9.2]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.3207, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.3, 95% CI 2-sided [-2.7 to 5.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0586, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.5, 95% CI 2-sided [-0.2 to 9.2]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0419, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.2, 95% CI 2-sided [0.3 to 10.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0244, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.3, 95% CI 2-sided [1.2 to 11.4]

9. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=50% Improvement (EASI-50) From Baseline at Weeks 2, 4, 8 and 12
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 35.7 [28.2 to 43.2] | 55.3 [47.4 to 63.2] | 10.5 [3.6 to 17.4]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 58.7 [51.0 to 66.5] | 78.4 [71.9 to 84.9] | 28.6 [18.5 to 38.7]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 66.2 [58.8 to 73.6] | 82.5 [76.5 to 88.5] | 34.6 [24.1 to 45.2]
  Week 12: number analyzed (Participants) | 155 | 154 | 77
  Week 12 | 68.4 [61.1 to 75.7] | 79.9 [73.5 to 86.2] | 19.5 [10.6 to 28.3]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 25.0, 95% CI 2-sided [14.8 to 35.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 44.2, 95% CI 2-sided [33.9 to 54.6]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 30.2, 95% CI 2-sided [17.5 to 42.8]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 49.8, 95% CI 2-sided [37.8 to 61.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 31.5, 95% CI 2-sided [18.8 to 44.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 47.6, 95% CI 2-sided [35.7 to 59.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 48.7, 95% CI 2-sided [37.2 to 60.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 60.1, 95% CI 2-sided [49.1 to 71.0]

10. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=90% Improvement (EASI-90) From Baseline at Weeks 2, 4, 8 and 12
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 2.5 [0.1 to 5.0] | 9.2 [4.6 to 13.8] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 9.7 [5.0 to 14.3] | 22.9 [16.2 to 29.5] | 0 [0.0 to 4.7]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 17.2 [11.3 to 23.1] | 34.4 [26.9 to 41.9] | 2.6 [0.0 to 6.1]
  Week 12: number analyzed (Participants) | 155 | 154 | 77
  Week 12 | 23.9 [17.2 to 30.6] | 37.7 [30.0 to 45.3] | 3.9 [0.0 to 8.2]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1623, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 2.5, 95% CI 2-sided [-1.7 to 6.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0070, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.1, 95% CI 2-sided [3.4 to 14.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0049, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.7, 95% CI 2-sided [4.0 to 15.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 22.9, 95% CI 2-sided [15.5 to 30.2]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 14.6, 95% CI 2-sided [7.2 to 22.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 31.6, 95% CI 2-sided [23.1 to 40.1]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.1, 95% CI 2-sided [11.9 to 28.3]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 33.5, 95% CI 2-sided [24.6 to 42.5]

11. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of 100% Improvement (EASI-100) From Baseline at Weeks 2, 4, 8 and 12
Description: EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 0 [0.0 to 2.3] | 1.3 [0.0 to 3.1] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 1.3 [0.0 to 3.1] | 3.9 [0.8 to 7.0] | 0 [0.0 to 4.7]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 1.3 [0.0 to 3.0] | 3.9 [0.8 to 7.0] | 0 [0.0 to 4.6]
  Week 12: number analyzed (Participants) | 155 | 154 | 77
  Week 12 | 5.2 [1.7 to 8.6] | 7.1 [3.1 to 11.2] | 0 [0.0 to 4.7]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; P-value could not be calculated since percentage of participants with events was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.7 to 3.7]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3261, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.3, 95% CI 2-sided [-2.8 to 5.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.3207, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.3, 95% CI 2-sided [-2.7 to 5.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0810, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 3.9, 95% CI 2-sided [-0.8 to 8.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.3207, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.3, 95% CI 2-sided [-2.7 to 5.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0810, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 3.8, 95% CI 2-sided [-0.7 to 8.4]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0419, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.2, 95% CI 2-sided [0.3 to 10.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0180, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 7.0, 95% CI 2-sided [1.8 to 12.2]

12. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 2, 4, 8 and 12
Description: as for outcome 11
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percent change
  Change at Week 2 | -39.2 [-43.8 to -34.7] | -51.3 [-55.9 to -46.7] | -9.0 [-15.4 to -2.5]
  Change at Week 4 | -54.3 [-59.1 to -49.5] | -69.0 [-73.7 to -64.2] | -24.4 [-31.1 to -17.7]
  Change at Week 8 | -59.5 [-65.0 to -54.0] | -73.2 [-78.7 to -67.7] | -33.0 [-41.1 to -25.0]
  Change at Week 12 | -60.0 [-66.5 to -53.6] | -73.3 [-79.7 to -66.9] | -28.6 [-38.4 to -18.8]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 2: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -30.2, 95% CI 2-sided [-38.1 to -22.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -42.3, 95% CI 2-sided [-50.3 to -34.4]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 4: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -29.9, 95% CI 2-sided [-38.1 to -21.7]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -44.6, 95% CI 2-sided [-52.8 to -36.3]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 8: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -26.4, 95% CI 2-sided [-36.2 to -16.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -40.2, 95% CI 2-sided [-50.0 to -30.4]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 12: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -31.4, 95% CI 2-sided [-43.1 to -19.7]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -44.7, 95% CI 2-sided [-56.4 to -33.0]

13. Secondary Outcome: Change From Baseline in the Percentage Body Surface Area (%BSA) Affected at Week 2, 4, 8, and 12
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of BSA
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of BSA
  Change at Week 2 | -27.8 [-33.0 to -22.6] | -35.4 [-40.6 to -30.2] | -1.3 [-8.7 to 6.0]
  Change at Week 4 | -45.0 [-50.4 to -39.6] | -55.7 [-61.1 to -50.3] | -15.3 [-22.9 to -7.7]
  Change at Week 8 | -53.4 [-60.0 to -46.8] | -61.1 [-67.7 to -54.5] | -20.5 [-30.1 to -10.9]
  Change at Week 12 | -56.4 [-63.1 to -49.6] | -65.0 [-71.7 to -58.3] | -16.8 [-26.9 to -6.6]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -26.5, 95% CI 2-sided [-35.5 to -17.5]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -34.1, 95% CI 2-sided [-43.1 to -25.1]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -29.7, 95% CI 2-sided [-39.0 to -20.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -40.5, 95% CI 2-sided [-49.8 to -31.1]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -32.9, 95% CI 2-sided [-44.6 to -21.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -40.6, 95% CI 2-sided [-52.2 to -28.9]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -39.6, 95% CI 2-sided [-51.8 to -27.4]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -48.2, 95% CI 2-sided [-60.4 to -36.0]

14. Secondary Outcome: Percentage of Participants With Percentage Body Surface Area (%BSA) (From EASI) < 5% at Weeks 2, 4, 8 and 12
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limb, 3.33% for trunk and 2.5% for lower limb. % BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 1.9 [0.0 to 4.1] | 5.9 [2.2 to 9.7] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 6.5 [2.6 to 10.3] | 17.0 [11.0 to 22.9] | 0 [0.0 to 4.7]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 15.9 [10.2 to 21.6] | 27.3 [20.2 to 34.3] | 1.3 [0.0 to 3.8]
  Week 12: number analyzed (Participants) | 155 | 154 | 77
  Week 12 | 22.6 [16.0 to 29.2] | 34.4 [26.9 to 41.9] | 3.9 [0.0 to 8.2]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2353, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.9, 95% CI 2-sided [-2.2 to 6.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0332, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.8, 95% CI 2-sided [0.8 to 10.8]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0227, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.5, 95% CI 2-sided [1.4 to 11.6]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 16.8, 95% CI 2-sided [10.1 to 23.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 14.5, 95% CI 2-sided [7.7 to 21.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 25.8, 95% CI 2-sided [18.1 to 33.4]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 18.5, 95% CI 2-sided [10.5 to 26.5]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 30.2, 95% CI 2-sided [21.4 to 39.0]

15. Secondary Outcome: Percentage of Participants Achieving Scoring Atopic Dermatitis (SCORAD) Response >=50% Improvement From Baseline at Week 2, 4, 8 and 12
Description: SCORAD: scoring index for AD combining extent, severity, subjective symptoms. Extent (A): rule of 9 was used to calculate BSA affected by AD as a % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. The score for each body region was added to determine A (0-100). Severity (B): severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none=0, mild=1, moderate=2,severe=3. The severity scores were summed to give B (0-18). Subjective symptoms (C): pruritus and sleep, each of these 2 were scored by participant/caregiver using visual analogue scale (VAS) where "0" = no itch/no sleeplessness and "10" = the worst imaginable itch/sleeplessness, higher scores=worse symptoms. Scores for itch and sleeplessness were added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD=worse outcome.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 12.7 [7.5 to 18.0] | 32.9 [25.4 to 40.4] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 36.1 [28.6 to 43.7] | 60.8 [53.0 to 68.5] | 7.8 [1.8 to 13.8]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 43.3 [35.6 to 51.1] | 61.7 [54.0 to 69.4] | 15.4 [7.4 to 23.4]
  Week 12: number analyzed (Participants) | 155 | 155 | 78
  Week 12 | 49.0 [41.2 to 56.9] | 62.6 [55.0 to 70.2] | 12.8 [5.4 to 20.2]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 12.7, 95% CI 2-sided [6.5 to 18.9]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 32.6, 95% CI 2-sided [24.6 to 40.6]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 28.3, 95% CI 2-sided [18.5 to 38.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 52.8, 95% CI 2-sided [43.2 to 62.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 28.0, 95% CI 2-sided [17.0 to 39.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 46.1, 95% CI 2-sided [35.2 to 57.1]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 36.2, 95% CI 2-sided [25.4 to 47.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 49.6, 95% CI 2-sided [38.9 to 60.3]

16. Secondary Outcome: Percentage of Participants Achieving Scoring Atopic Dermatitis (SCORAD) Response >=75% Improvement From Baseline at Week 2, 4, 8 and 12
Description: SCORAD: scoring index for AD combining extent, severity, subjective symptoms. Extent (A): rule of 9 was used to calculate BSA affected by AD as a % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. The score for each body region was added to determine A (0-100). Severity (B): severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none (0), mild (1), moderate (2) or severe (3). The severity scores added to give B (0-18). Subjective symptoms (C): pruritus and sleep loss, each of these 2 were scored by participant/caregiver using VAS where "0" = no itch or no sleeplessness and "10" = the worst imaginable itch or sleeplessness, higher scores worse symptoms. Scores for itch and sleeplessness added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD = worse outcome.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percentage of participants
  Week 2: number analyzed (Participants) | 157 | 152 | 76
  Week 2 | 1.9 [0.0 to 4.1] | 5.3 [1.7 to 8.8] | 0 [0.0 to 4.7]
  Week 4: number analyzed (Participants) | 155 | 153 | 77
  Week 4 | 7.1 [3.1 to 11.1] | 17.6 [11.6 to 23.7] | 0 [0.0 to 4.7]
  Week 8: number analyzed (Participants) | 157 | 154 | 78
  Week 8 | 11.5 [6.5 to 16.4] | 26.0 [19.0 to 32.9] | 0 [0.0 to 4.6]
  Week 12: number analyzed (Participants) | 155 | 155 | 78
  Week 12 | 18.7 [12.6 to 24.8] | 30.3 [23.1 to 37.6] | 2.6 [0.0 to 6.1]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2261, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.9, 95% CI 2-sided [-2.2 to 6.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0451, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.2, 95% CI 2-sided [0.3 to 10.0]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.0171, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 7.0, 95% CI 2-sided [1.8 to 12.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 17.7, 95% CI 2-sided [10.9 to 24.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.0018, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 11.5, 95% CI 2-sided [5.5 to 17.5]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 25.7, 95% CI 2-sided [18.3 to 33.1]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 16.2, 95% CI 2-sided [8.8 to 23.6]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 27.6, 95% CI 2-sided [19.3 to 35.8]

17. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Visual Analogue Scale (VAS) of Itch at Weeks 2, 4, 8 and 12
Description: as for outcome 16
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
units on a scale
  Change at Week 2 | -2.3 [-2.7 to -2.0] | -3.5 [-3.8 to -3.1] | -0.6 [-1.1 to -0.1]
  Change at Week 4 | -3.1 [-3.5 to -2.7] | -4.3 [-4.6 to -3.9] | -1.2 [-1.7 to -0.6]
  Change at Week 8 | -3.4 [-3.8 to -3.0] | -4.3 [-4.7 to -4.0] | -1.8 [-2.4 to -1.2]
  Change at Week 12 | -3.5 [-3.9 to -3.1] | -4.2 [-4.7 to -3.8] | -2.1 [-2.7 to -1.4]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Week 2: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category), baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.7, 95% CI 2-sided [-2.3 to -1.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.9, 95% CI 2-sided [-3.5 to -2.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; Week 4: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category), baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.9, 95% CI 2-sided [-2.6 to -1.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -3.1, 95% CI 2-sided [-3.8 to -2.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; Week 8: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category), baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.6, 95% CI 2-sided [-2.3 to -0.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.6, 95% CI 2-sided [-3.3 to -1.9]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; Week 12: MMRM contained fixed factors of treatment, visit, treatment by visit interaction, randomization strata (baseline disease severity and age category), baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Difference in LS mean = -1.4, 95% CI 2-sided [-2.2 to -0.6]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.2, 95% CI 2-sided [-3.0 to -1.4]

18. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Visual Analogue Scale (VAS) Sleep Loss at Weeks 2, 4, 8 and 12
Description: as for outcome 16
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
units on a scale
  Change at Week 2 | -1.9 [-2.2 to -1.5] | -2.9 [-3.3 to -2.5] | -0.5 [-1.0 to 0.0]
  Change at Week 4 | -2.8 [-3.1 to -2.4] | -3.9 [-4.3 to -3.6] | -1.0 [-1.5 to -0.5]
  Change at Week 8 | -3.1 [-3.5 to -2.7] | -3.9 [-4.3 to -3.5] | -1.5 [-2.1 to -0.9]
  Change at Week 12 | -3.0 [-3.4 to -2.6] | -3.8 [-4.2 to -3.4] | -2.1 [-2.7 to -1.5]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.4, 95% CI 2-sided [-2.0 to -0.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.4, 95% CI 2-sided [-3.0 to -1.8]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 17, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.8, 95% CI 2-sided [-2.4 to -1.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -3.0, 95% CI 2-sided [-3.6 to -2.3]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.6, 95% CI 2-sided [-2.3 to -0.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.4, 95% CI 2-sided [-3.1 to -1.7]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 17, analysis 7]; Test type: Superiority; p = 0.0164, Mixed Models Analysis; Difference in LS mean = -0.9, 95% CI 2-sided [-1.7 to -0.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 17, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.7, 95% CI 2-sided [-2.5 to -1.0]

19. Secondary Outcome: Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Total Score at Week 2, 4, 8 and 12
Description: as for outcome 16
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 158 | 155 | 78
percent change
  Change at Week 2 | -27.2 [-30.5 to -23.9] | -38.5 [-41.8 to -35.1] | -6.3 [-11.0 to -1.6]
  Change at Week 4 | -38.9 [-42.6 to -35.1] | -53.1 [-56.9 to -49.4] | -17.2 [-22.5 to -12.0]
  Change at Week 8 | -42.6 [-46.7 to -38.4] | -56.7 [-60.9 to -52.6] | -23.1 [-29.2 to -17.1]
  Change at Week 12 | -45.8 [-50.9 to -40.7] | -56.2 [-61.2 to -51.1] | -22.7 [-30.4 to -15.1]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -20.9, 95% CI 2-sided [-26.6 to -15.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -32.1, 95% CI 2-sided [-37.9 to -26.4]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -21.6, 95% CI 2-sided [-28.1 to -15.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -35.9, 95% CI 2-sided [-42.3 to -29.4]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -19.4, 95% CI 2-sided [-26.8 to -12.1]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -33.6, 95% CI 2-sided [-41.0 to -26.3]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -23.1, 95% CI 2-sided [-32.3 to -13.9]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -33.4, 95% CI 2-sided [-42.6 to -24.3]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study.
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/158 | 0/155 | 0/78
Serious Adverse Events (participants affected / at risk) | 5/158 | 2/155 | 1/78
Other Adverse Events (participants affected / at risk) | 56/158 | 52/155 | 22/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 100 mg (N=158) | PF-04965842 200 mg (N=155) | Placebo (N=78)
Sudden death (General disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 1
Herpangina (Infections and infestations) | 1 | 0 | 0
Osteomyelitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 100 mg (N=158) | PF-04965842 200 mg (N=155) | Placebo (N=78)
Nausea (Gastrointestinal disorders) | 12 | 22 | 2
Vomiting (Gastrointestinal disorders) | 2 | 8 | 1
Nasopharyngitis (Infections and infestations) | 20 | 12 | 5
Upper respiratory tract infection (Infections and infestations) | 14 | 5 | 3
Headache (Nervous system disorders) | 9 | 12 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 9 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9 | 6 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03575871/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT03575871/SAP_001.pdf